CLINICAL TRIAL: NCT05046262
Title: Calcium Electroporation for Basal Cell Carcinomas - Proof of Concept Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Mirai Medical, Ireland (Unknown)
Responsible Party: Principal Investigator, Stine Wiegell, MD, PhD, DMSc, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2019-002730-36
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Calcium Chloride; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Calcium chloride — Calcium electroporation
  Other Names: electroporation

SUMMARY:
25 patients with primary low-risk basal cell carcinoma treated with calcium electroporation

DETAILED DESCRIPTION:
25 patients with primary low-risk basal cell carcinoma treated with calcium electroporation, if partial or no response after 3 months the treatment was repeated. Follow-up 3 and 12 months after last treatment.

ELIGIBILITY:
Inclusion Criteria:

Primary low risk basal cell carcinoma less than 3 cm in diameter

-

Exclusion Criteria:

Immunosuppression or organ transplant recipients Pregnancy or breastfeeding Allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-02-22 (Estimated); Study Completion 2022-02-22 (Estimated)

PRIMARY OUTCOMES:
complete response | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided